CLINICAL TRIAL: NCT00681538
Title: A Two-phase, Phase 3 Study of the Safety and Efficacy of Sativex, in the Symptomatic Relief of Spasticity in Subjects With Spasticity Due to Multiple Sclerosis: Phase A - Single-blind Response Assessment; Phase B - Double-blind, Randomised, Placebo Controlled, Parallel Group Study.
Brief Title: A Study of the Safety and Effectiveness of Sativex®, for the Relief of Symptoms of Spasticity in Subjects, From Phase B, With Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GWSP0604
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2011-12-07 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Spasticity; Multiple Sclerosis
Keywords: Spasticity; Multiple Sclerosis
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental): Contains Δ9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml, as extracts of Cannabis sativa L.
  Subjects received study medication delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 12 actuations (THC 32.4 mg:CBD 30 mg) in 24 hours
  Interventions: Drug: Sativex®
- Placebo (Placebo Comparator): Contains no active drug but colourants and excipients. Subjects received placebo delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 12 actuations in 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex® — containing THC (27 mg/ml):CBD (25 mg/ml), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Maximum dose within any 24-hour interval is 12 sprays (THC 32.4 mg: CBD 30 mg)
  Other Names: GW-1000-02
  Arms: Sativex
Drug: Placebo — containing ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring and colouring FD&C Yellow No.5 (E102 tartrazine) (0.0260%), FD&C Yellow No.6 (E110 sunset yellow) (0.0038%), FD&C Red No. 40 (E129 Allura red AC) (0.00330%) and FD&C Blue No.1 (E133 Brilliant blue FCF) (0.00058%).
  Other Names: GA0034
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Sativex® versus Placebo is effective in the relief of symptoms of spasticity in subjects with multiple sclerosis, who have been identified as having a capacity to respond to Sativex.

DETAILED DESCRIPTION:
This 19 week, multicentre study was conducted in two phases. Phase A was a preliminary, single-blind four week treatment period to identify subjects with a capacity to respond to Sativex; eligible, consenting subjects entered a seven day screening period prior to returning to the study centre to begin a four week single-blind course of Sativex treatment. At the end of this phase, subjects' response to Sativex was assessed; those with the capacity to respond (i.e. at least a 20% reduction in mean 0-10 point numerical rating scale (NRS) spasticity score between screening and the end of the four week Phase A treatment) were eligible for entry into Phase B while those who did not respond took no further part in the study other than a follow up visit 14 days later.

Phase B was a 12 week double-blind, randomised, placebo controlled, parallel group study with visits at 28 day intervals and a final follow up visit 14 days after completion or withdrawal.

The level of spasticity, spasm frequency and sleep disruption were collected each day during the entire study via an interactive voice response system (IVRS). In addition, study medication dosing data were recorded via IVRS throughout Phases A and B. Assessments of other secondary and functional measures of spasticity, safety and tolerability, QOL (quality of life) and mood were also gathered throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the study.
* Male or female, aged 18 years or above.
* Subject is able (in the investigator's opinion) and willing to comply with all study requirements.
* Diagnosed with any disease sub-type of MS of at least six months duration.
* Spasticity due to MS of at least three months duration, which is not wholly relieved with current anti-spasticity therapy, and which is expected to remain stable for the duration of the study.
* Subject fulfils at least one of the two criteria below. Subject must be either: Currently established on a regular dose of anti-spasticity therapy or Previously tried and failed, or could not tolerate suitable anti-spasticity therapy.
* Subject is currently receiving a stable regimen (for at least 30 days prior to study entry) of all medications that may have an effect on spasticity; and willing to maintain this for the duration of the study. If the subject is currently taking disease-modifying medication, this must be at a stable dose for at least three months prior to the screening visit; the dose must also remain stable for the duration of the study.
* Willing for his or her name to be notified to his or her primary care physician, and consultant and the responsible authorities for participation in this study, as applicable.

Exclusion Criteria:

* Any concomitant disease or disorder that has spasticity-like symptoms or that may influence the subject's level of spasticity.
* Subject's medical history suggests that relapse/remission is likely to occur during the study (over the next 19 weeks) which, in the opinion of the investigator, is expected to influence the subject's spasticity.
* Currently receiving a prohibited medication and unwilling to stop for the stated period prior to the screening visit and for the duration of the study.
* Any known or suspected history of: schizophrenia or other psychotic illness;diagnosed dependence disorder;poorly controlled epilepsy or recurrent seizures;hypersensitivity to cannabinoids.
* Significant cardiac, renal or hepatic disease.
* Female subjects of child bearing potential and male subjects whose partner is of child bearing potential, unless willing to ensure that they or their partner use effective contraception during the study and for three months thereafter.
* Female subject who is pregnant, lactating or planning pregnancy during the course of the study or for three months thereafter.
* Subjects who have received an IMP within the 12 weeks before Visit 1.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the result of the study, or the subject's ability to participate in the study.
* Following a physical examination, the subject has any abnormalities that, in the opinion of the investigator, would prevent them from safely participating in the study.
* Unwilling to abstain from donation of blood during the study.
* Travel outside the country of residence planned during the study.
* Subjects previously randomised into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Davies, MRCP, FRCP, Principal Investigator — Department of Neurology
Locations (1):
- Department of Neurology, Northampton General Hospital, Cliftonville, Northampton, United Kingdom

REFERENCES:
- [Result] Novotna A, Mares J, Ratcliffe S, Novakova I, Vachova M, Zapletalova O, Gasperini C, Pozzilli C, Cefaro L, Comi G, Rossi P, Ambler Z, Stelmasiak Z, Erdmann A, Montalban X, Klimek A, Davies P; Sativex Spasticity Study Group. A randomized, double-blind, placebo-controlled, parallel-group, enriched-design study of nabiximols* (Sativex((R)) ), as add-on therapy, in subjects with refractory spasticity caused by multiple sclerosis. Eur J Neurol. 2011 Sep;18(9):1122-31. doi: 10.1111/j.1468-1331.2010.03328.x. Epub 2011 Mar 1. PMID 21362108

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only those subjects who were deemed responders to Sativex from Phase A (i.e. at least a 20% reduction in mean 0-10 point numerical rating scale (NRS) spasticity score between screening and the end of the four week Phase A treatment) were eligible to enter Phase B of the study.
Groups:
- Sativex (Phase B): contains Δ9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml, as extracts of Cannabis sativa L.Subjects received study medication delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 12 actuations (THC 32.4 mg:CBD 30 mg) in 24 hours.
- Placebo (Phase B): Contains no active drug but colourants and excipients. Subjects received placebo delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 12 actuations in 24 hours.
Period: Phase A- 4 Weeks Single Blind
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Started | 572 | 0
Completed | 538 | 0
Not Completed | 34 | 0
Period: Phase B- Responders;12 Week Double-blind
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Started | 124 | 117
Completed | 109 | 115
Not Completed | 15 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex (Phase B) | Placebo (Phase B) | Total
Number analyzed (Participants) | 124 | 117 | 241
Age, Continuous [Mean (Standard Deviation); unit: Years] — Of the 572 subjects who entered Phase A, 241 entered Phase B; 124 randomised to Sativex and 117 to placebo. The data below details that for Phase B.
  Years | 49.1 (9.09) | 48.1 (9.59) | 48.6 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 73 | 145
  Male | 52 | 44 | 96
Duration of Multiple Sclerosis Phase B [Mean (Standard Deviation); unit: years] — Of the 572 subjects who entered Phase A, 241 entered Phase B; 124 randomised to Sativex and 117 to placebo.
  years | 13.3 (8.29) | 11.8 (7.38) | 12.6 (7.88)
Duration of Spasticity Phase B [Mean (Standard Deviation); unit: years] — Of the 572 subjects who entered Phase A, 241 entered Phase B; 124 randomised to Sativex and 117 to placebo.
  years | 8.6 (6.89) | 6.7 (5.40) | 7.7 (6.27)
Expanded Disability Status Scale (EDSS)- Phase B [Mean (Standard Deviation); unit: Score] — 241 entered Phase B; 124 randomised to Sativex and 117 to placebo. EDSS is a method of quantifying disability in multiple sclerosis.The EDSS quantifies disability in eight Functional Systems (FS) and allows neurologists to assign a Functional System Score in each of these. EDSS steps 1.0 to 4.5 refer to people with MS who are fully ambulatory. EDSS steps 5.0 to 9.5 are defined by the impairment to ambulation. Each score is given a definition and thus can identify for the subject their score depending on their condition e.g. score of 1.0: No disability, minimal signs on 1 FS.
  Score | 6.5 (1.46) | 6.0 (1.44) | 6.0 (1.45)
Baseline Spasticity numerical rating scale (NRS) Score Phase B [Mean (Standard Deviation); unit: Score] — Of the 572 subjects who entered Phase A, 241 entered Phase B; 124 randomised to Sativex and 117 to placebo.
  Subjects were asked "On a scale of '0 to 10' please indicate the average level of your spasticity over the last 24 hours" with the anchors: 0 = 'no spasticity' and 10 = 'worst possible spasticity'. They were asked to relate 'no spasticity' to the time prior to the onset of their spasticity.
  Score | 3.87 (1.49) | 3.92 (1.55) | 3.90 (1.51)

OUTCOME MEASURES:

1. Primary Outcome: The Change in Mean Spasticity Numerical Rating Scale (NRS) Score From Baseline to End of Treatment (Phase B).
Description: Subjects were asked "On a scale of '0 to 10' please indicate the average level of your spasticity over the last 24 hours" with the anchors: 0 = 'no spasticity' and 10 = 'worst possible spasticity'. They were asked to relate 'no spasticity' to the time prior to the onset of their spasticity.
Time Frame: Baseline (last 7 days of Week 4) - End of treatment (last 7 days of Week 17)
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 124 | 117
Points on scale | 3.68 (1.83) | 4.56 (2.31)
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p = 0.0002, ANCOVA; Treatment Difference = -0.84, 95% CI 2-sided [-1.29 to -0.40]

2. Secondary Outcome: Number of Subjects Showing an Improvement of at Least 30% or 50% in Their Mean NRS Spasticity Score (Phase B) From Baseline.
Description: A subject was classified as a responder in the evaluable period provided they did not withdraw due to lack of efficacy and achieved at least a 30% or 50% reduction (i.e. improvement) in the mean NRS spasticity score from baseline (Day 1) to the end of treatment(last 7 days of Week 17 Phase B). All other subjects and subjects without evaluable data were considered non-responders.
Time Frame: Baseline (Day 1) - End of treatment (last 7 days of Week 17)
Measure: Number; unit: participants
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 124 | 117
participants
  30% improvement in spasticity | 92 | 60
  50% improvement in spasticity | 56 | 39
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); 30% responders; Test type: Superiority or Other; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 2.731, 95% CI 2-sided [1.589 to 4.694] — Odds ratio>1 indicates an improvement in favour of Sativex
Statistical Analysis 2: Comparison: Sativex (Phase B) vs Placebo (Phase B); 50% Responders; Test type: Superiority or Other; p = 0.0612, Regression, Logistic; Odds Ratio (OR) = 1.647, 95% CI 2-sided [0.977 to 2.777] — Odds ratio>1 indicates an improvement in favour of Sativex

3. Secondary Outcome: Change in Spasm Frequency (Number of Spasms Per Day) From Baseline to End of Treatment (Phase B).
Description: The subjects' baseline spasm frequency was the mean of the last seven days scores (Week 4) of Phase A treatment. The variable for analysis was the change in mean spasm frequency from baseline to the end of treatment (last 7 days of Week 17 Phase B).
Time Frame: Baseline (last 7 days of Week 4) - End of treatment (last 7 days of Week 17)
Measure: Mean (Standard Deviation); unit: Spasms per day
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 124 | 117
Spasms per day | 5.56 (10.33) | 7.70 (12.02)
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p = 0.0046, ANCOVA; Treatment difference = -2.53, 95% CI 2-sided [-4.27 to -0.79] — A negative difference indicates an improvement in spasm frequency in favour of Sativex

4. Secondary Outcome: Change in Sleep Disruption (Daily 11-point NRS) From Baseline to End of Treatment (Phase B).
Description: The sleep disruption NRS score was recorded by subjects via a daily call to the interactive voice response system at bedtime. Subjects were asked "On a scale of '0 to 10' please indicate how you your spasticity disrupted your sleep last night" with the anchors: 0 = 'did not disrupt sleep' and 10 = 'completely disrupted (unable to sleep at all)'.
Time Frame: Baseline (last 7 days of Week 4) - End of treatment (last 7 days of Week 17)
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 124 | 117
Points on scale | 1.71 (1.65) | 2.65 (2.45)
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p < 0.0001, ANCOVA; treatment difference = -0.88, 95% CI 2-sided [-1.25 to -0.51] — A negative difference indicates an improvement in sleep disruption in favour of Sativex

5. Secondary Outcome: Change in Spasticity as Measured Using the Modified Ashworth Scale From Baseline to End of Treatment (Phase B).
Description: All 20 muscle groups were assessed for spasticity (using a 1-5 scale): 1= no increase in muscle tone to 5= passive movement is difficult and affected part is rigid in flexion or extension. The score for all 20 muscle groups were added to give a total score out of 100; minimum score was 20. A decrease in score indicates an improvement in condition.
Time Frame: Baseline (End of Week 4) - End of treatment (End of Week 17)
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 121 | 116
Score on scale | -0.1 (8.25) | 1.8 (7.79)
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p = 0.0939, ANCOVA; treatment difference = -1.75, 95% CI 2-sided [-3.80 to 0.30] — A negative difference indicates an improvement in spasticity in favour of Sativex

6. Secondary Outcome: Change in Motricity Index Score From Baseline to End of Treatment (Phase B)for Affected Limbs.
Description: Arm - 3 movements were pinch grip, elbow flexion and shoulder abduction. Leg - 3 movements were ankle dorsiflexion, knee extension and hip flexion. The total arm and leg score was the addition of the score for the 3 arm movements and 3 leg movements, respectively. One point was then added to each limb score to give a maximum score of 100; minimum was 1 point. Where both arms (or both legs) were assessed, the average of the two limbs scores was used as the assessment score; otherwise the affected limb total score was used. An increase in score indicates an improvement in condition.
Time Frame: Baseline (End of Week 4) - End of treatment (End of Week 17)
Population: For Arm subject numbers were 23 for Sativex and 22 for placebo. For Leg subject numbers were 91 for Sativex and 92 for placebo.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 124 | 117
Score on scale
  Arm | 0.5 (15.62) | 0.8 (10.60)
  Leg | -1.3 (7.64) | -1.0 (9.48)
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); For Arm; Test type: Superiority or Other; p = 0.56, ANCOVA; treatment difference = -2.85, 95% CI 2-sided [-12.75 to 7.04] — A positive treatment difference indicates an improvement in favour of Sativex
Statistical Analysis 2: Comparison: Sativex (Phase B) vs Placebo (Phase B); For leg; Test type: Superiority or Other; p = 0.98, ANCOVA; Treatment difference = 0.04, 95% CI 2-sided [-2.56 to 2.64] — A positive treatment difference indicates an improvement in favour of Sativex

7. Secondary Outcome: Change in Timed 10-metre Walk From Baseline to End of Treatment (Phase B).
Description: Only those subjects for whom it was appropriate (i.e. ambulatory subjects) were timed how long it took to walk 10 metres. Walk time was only assessed for subjects who successfully completed the Timed 10 Metre Walk. A negative difference from baseline indicates an improvement walk time.
Time Frame: Baseline (End of Week 4) - End of treatment (End of Week 17)
Population: Only those subjects for whom it was appropriate (i.e. ambulatory subjects) were timed how long it took to walk 10 metres. Walk time was only assessed for subjects who successfully completed the Timed 10 Metre Walk.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 84 | 83
Seconds | -2.3 (8.38) | 2.0 (15.16)
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p = 0.0687, ANCOVA; Treatment difference = -3.34, 95% CI 2-sided [-6.95 to 0.26] — A negative treatment difference indicates an improvement in favour of Sativex

8. Secondary Outcome: Subject Global Impressions of Change at End of Treatment (Phase B).
Time Frame: End of Treatment (WeeK 17)
Measure: Number; unit: participants
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 121 | 117
participants
  Very much better | 14 | 10
  Much better | 40 | 28
  Minimally better | 39 | 33
  No change | 17 | 35
  Minimally worse | 4 | 7
  Much worse | 6 | 1
  Very much worse | 1 | 3
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p = 0.0234, Regression, Logistic; Odds Ratio (OR) = 1.703, 95% CI 2-sided [1.075 to 2.698] — An odds ratio > 1 indicates an improvement in favour of Sativex

9. Secondary Outcome: Carer Global Impressions of Change at of Treatment (Phase B).
Time Frame: End of treatment (Week 17)
Population: Sample sizes were reduced as not all subjects had a Carer to make this assessment.
Measure: Number; unit: participants
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 71 | 69
participants
  Very much better | 2 | 0
  Much better | 15 | 11
  Minimally better | 31 | 19
  No change | 16 | 24
  Minimally worse | 4 | 8
  Much worse | 2 | 5
  Very much worse | 1 | 2
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p = 0.0053, Regression, Logistic; Odds Ratio (OR) = 2.400, 95% CI 2-sided [1.297 to 4.443] — An odds ratio > 1 indicates an improvement in favour of Sativex

10. Secondary Outcome: Carer Ease of Transfer Global Impressions of Change at End of Treatment (Phase B).
Time Frame: End of treatment (week 17)
Population: Sample sizes were reduced as not all subjects had a Carer to make this assessment.
Measure: Number; unit: participants
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 71 | 69
participants
  Very much better | 1 | 1
  Much better | 9 | 8
  Minimally better | 27 | 14
  No change | 24 | 30
  Minimally worse | 6 | 11
  Much worse | 4 | 3
  Very much worse | 0 | 2
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p = 0.0613, Regression, Logistic; Odds Ratio (OR) = 1.792, 95% CI 2-sided [0.973 to 3.301] — An odds ratio > 1 indicates an improvement in favour of Sativex

11. Secondary Outcome: Physician Global Impressions of Change at End of Treatment (Phase B).
Time Frame: End of treatment (week 17)
Measure: Number; unit: participants
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 122 | 117
participants
  Very much better | 6 | 8
  Much better | 44 | 29
  Minimally better | 45 | 26
  No change | 17 | 37
  Minimally worse | 4 | 13
  Much worse | 6 | 4
  Very much worse | 0 | 0
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p = 0.0045, Regression, Logistic; Odds Ratio (OR) = 1.958, 95% CI 2-sided [1.232 to 3.112] — An odds ratio > 1 indicates an improvement in favour of Sativex

12. Secondary Outcome: Change EuroQoL Quality of Life Questionnaire (EQ-5D)From Baseline to End of Treatment (Phase B)
Description: The EQ-5D questionnaire provided two outcomes:
  1. A weighted health state index visual analogue scale (VAS)
  2. A self-rated health status VAS EQ-5D Health Status VAS Scale: 0 = worst health state imaginable to 100 = best health state imaginable. An increase in score indicates an improvement in condition.
  The weighted health state index used the same VAS as above but was calculated for each assessment without imputation to account for missing values i.e., if one or more individual items was missing then the whole index was missing.
Time Frame: [Baseline (End of Week 4) - End of treatment (End of Week 17)
Population: EQ-5D Health State Index Sativex n=117 and placebo n=111. EQ-5D Health Status VAS Sativex n=121 and placebo n=117.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 124 | 117
score on scale
  EQ-5D Health State Index | 0.003 (0.155) | -0.013 (0.176)
  EQ-5D Health Status VAS | -0.7 (15.3) | -2.8 (19.9)
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); For Health State Index; Test type: Superiority or Other; p = 0.2836, ANCOVA; Treatment Difference = 0.02, 95% CI 2-sided [-0.02 to 0.07] — A positive difference indicates an improvement in favour of Sativex
Statistical Analysis 2: Comparison: Sativex (Phase B) vs Placebo (Phase B); Health Status VAS; Test type: Superiority or Other; p = 0.5644, ANCOVA; Treatment Difference = 1.24, 95% CI 2-sided [-3.01 to 5.50] — A positive difference indicates an improvement in favour of Sativex

13. Secondary Outcome: Mood Assessment: Change in Beck Depression Inventory - II (BDI-II)From Baseline to End of Treatment (Phase B)
Description: This was a 21-question multiple choice self-report inventory. Subjects' responses to the 21 questions were assigned a score ranging from zero to three, indicating the severity of the symptom. The sum of all BDI-II question scores indicated the severity of depression; score range 0-63. An decrease in score indicates an improvement in condition.
Time Frame: Baseline (End of week 4) - end of treatment (end of week 17)
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Number analyzed (Participants) | 114 | 113
Score on scale | 0.5 (5.01) | 0.4 (6.54)
Statistical Analysis 1: Comparison: Sativex (Phase B) vs Placebo (Phase B); Test type: Superiority or Other; p = 0.9369, ANCOVA; Treatment Difference = -0.06, 95% CI 2-sided [-1.62 to 1.49] — A negative difference indicates an improvement in depression in favour of Sativex

ADVERSE EVENTS:
Time Frame: All AEs occurring from Baseline(week 4) to end of treatment (Week 17) (Phase B) i.e. 13 weeks were collected. All deaths and SAEs occurring within 28 days of the final dose of study medication were also collected.
Description: All AEs occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex (Phase B) | Placebo (Phase B)
Serious Adverse Events (participants affected / at risk) | 6/124 | 1/117
Other Adverse Events (participants affected / at risk) | 66/124 | 40/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (Phase B) (N=124) | Placebo (Phase B) (N=117)
Bronchopneumonia (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
MS Relapse (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (Phase B) (N=124) | Placebo (Phase B) (N=117)
Urinary tract infection (Infections and infestations) | 9 | 12
Nasopharyngitis (Infections and infestations) | 4 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 5
Headache (Nervous system disorders) | 2 | 5
Muscle spasticity (Nervous system disorders) | 3 | 4
Somnolence (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 4 | 0
MS relapse (Nervous system disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 6
Dry mouth (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 6 | 1
Euphoric mood (Psychiatric disorders) | 4 | 1
Vertigo (Ear and labyrinth disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications for example, manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.